CLINICAL TRIAL: NCT02637063
Title: Interactive Web Program and Health Coaching for Prehypertensive Adults
Acronym: Prehype
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Center for Applied Science, Inc. (Industry)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R44HL095229 (NIH); R44HL095229 (NIH)
Record Dates: First submitted 2015-11-09; First posted 2015-12-22 (Estimated); Results first posted 2017-03-15 (Actual); Last update posted 2017-03-15 (Actual); Status verified 2017-01

CONDITIONS: Weight; Blood Pressure
Keywords: Lifestyle behavior change
MeSH Terms: conditions — Body Weight

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- BlipHub mobile-web app (Experimental): Mobile web app to promote blood-pressure-reducing diet, physical activity and weight loss.
  Interventions: Behavioral: BlipHub mobile-web app
- BlipHub mobile-web app + health coaching (Experimental): Telephonic coach-supported mobile web app to promote blood-pressure-reducing diet, physical activity and weight loss.
  Interventions: Behavioral: BlipHub mobile-web app + health coaching
- Usual care (Other): No intervention beyond the participants' personal medical care.
  Interventions: Other: Usual care

INTERVENTIONS:
Behavioral: BlipHub mobile-web app — Mobile web app to promote blood-pressure-reducing diet, physical activity and weight loss.
  Arms: BlipHub mobile-web app
Behavioral: BlipHub mobile-web app + health coaching — Telephonic coach-supported mobile web app to promote blood-pressure-reducing diet, physical activity and weight loss.
  Arms: BlipHub mobile-web app + health coaching
Other: Usual care — No intervention beyond participants' own medical care.
  Arms: Usual care

SUMMARY:
This project will develop and evaluate an interactive blood pressure self-management program for adults with prehypertension. The program will target blood pressure self-monitoring and the five proven lifestyle modifications recommended by JNC-7: weight reduction, the Dietary Approaches to Stop Hypertension (DASH) diet, sodium reduction, physical activity, and alcohol consumption.

The multi-modal program uses a combination of brief motivational health coaching, periodic engagement emails, and a robust interactive website to motivate people to take charge of their blood pressure management before they require medication. All program components were designed to conform to the underlying principles of motivational interviewing. Key program components include the use of email and Web-based social networking, personal stories, and a brief motivational coaching session to engage participants and encourage intrinsically motivated behavior changes. Self-assessment and tracking tools are combined with educational content to help participants align their daily lifestyle choices with their personal goals.

The Phase I prototype program promoted moderate physical activity and eating fruits and vegetables as part of the DASH diet. Results from the within-group (n = 39) evaluation showed moderate-to-large effect sizes for pre-to-post change in motivation, preparation behavior, self-efficacy, attitudes, and knowledge, and a small significant increase in physical activity. Participants gave the online program high ratings on satisfaction and usability, and reported improvements in confidence, readiness, clarity, change strategies, and interest in visiting the Website as a result of the coaching session.

The fully developed Phase II product will be evaluated in a large randomized trial (N = 450) with a 3-month intensive intervention, a 3-month maintenance intervention, and a 3-month follow-up period. The Phase II trial is expected to show reductions in blood pressure and improvements in JNC-recommended health behaviors. These changes in the outcome measures are expected to be mediated by changes in knowledge, attitudes, self-efficacy, behavioral intention, motivation, and patient activation.

DETAILED DESCRIPTION:
Approximately a third (31%) of adult Americans are prehypertensive (SBP 120-139 and/or DBP 80-89). Health care providers struggle to provide effective support for blood-pressure-lowering behavior changes, while patients continue to progress to full hypertension and the use of antihypertensive medications. Insurers and providers with access to electronic medical records, claims, and other medical data are in a unique position to identify prehypertensive adults and target them with a blood pressure self-management program. Preventing or delaying hypertension should reduce mid-term costs of antihypertensive medications and, more importantly, long-term costs of care for heart disease and stroke.

This project will develop and evaluate an interactive blood pressure self-management program for adults with prehypertension. The program will target blood pressure self-monitoring and the five proven lifestyle modifications recommended by JNC-7: weight reduction, the Dietary Approaches to Stop Hypertension (DASH) diet, sodium reduction, physical activity, and alcohol consumption.

The multi-modal program uses a combination of brief motivational health coaching, periodic engagement emails, and a robust interactive website to motivate people to take charge of their blood pressure management before they require medication. All program components were designed to conform to the underlying principles of motivational interviewing. Key program components include the use of email and Web-based social networking, personal stories, and a brief motivational coaching session to engage participants and encourage intrinsically motivated behavior changes. Self-assessment and tracking tools are combined with educational content to help participants align their daily lifestyle choices with their personal goals.

The Phase I prototype program promoted moderate physical activity and eating fruits and vegetables as part of the DASH diet. Results from the within-group (n = 39) evaluation showed moderate-to-large effect sizes for pre-to-post change in motivation, preparation behavior, self-efficacy, attitudes, and knowledge, and a small significant increase in physical activity. Participants gave the online program high ratings on satisfaction and usability, and reported improvements in confidence, readiness, clarity, change strategies, and interest in visiting the Website as a result of the coaching session.

The fully developed Phase II product will be evaluated in a large randomized trial (N = 450) with a 3-month intensive intervention, a 3-month maintenance intervention, and a 3-month follow-up period. The Phase II trial is expected to show reductions in blood pressure and improvements in JNC-recommended health behaviors. These changes in the outcome measures are expected to be mediated by changes in knowledge, attitudes, self-efficacy, behavioral intention, motivation, and patient activation.

ELIGIBILITY:
Inclusion Criteria

* Blood pressure in the JNC-7-defined prehypertension range (SBP 120-139 and/or DBP 80-89)
* Must be at least 18 years old
* Must be employed at least part time
* Must have access to the internet through a WIFI connection in a place where subject was willing to take BP and weight measurements
* Must be the only participant per household in the study

Exclusion Criteria

* Female subjects must not be pregnant or planning to get pregnant over the course of study
* Must not have experienced a stroke, heart attack, or heart disease diagnosis in the prior six months
* Must not be taking antihypertensive medications for any reason

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 203 (Actual)
Dates: Start 2013-11; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amelia J. Birney, MPH, MCHES, Principal Investigator — Oregon Center for Applied Science, Inc.
Locations (1):
- ORCAS, Eugene, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | BlipHub Mobile-web App | BlipHub Mobile-web App + Health Coaching | Usual Care
Started | 67 | 68 | 68
Completed | 62 | 64 | 62
Not Completed | 5 | 4 | 6
Not completed — Lost to Follow-up | 3 | 2 | 3
Not completed — Withdrawal by Subject | 2 | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BlipHub Mobile-web App | BlipHub Mobile-web App + Health Coaching | Usual Care | Total
Number analyzed (Participants) | 67 | 68 | 68 | 203
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 67 | 68 | 68 | 203
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 43 | 45 | 129
  Male | 26 | 25 | 23 | 74
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 9 | 6 | 19
  Not Hispanic or Latino | 63 | 59 | 62 | 184
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 1 | 3
  Asian | 3 | 2 | 2 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 12 | 11 | 12 | 35
  White | 46 | 48 | 47 | 141
  More than one race | 3 | 1 | 3 | 7
  Unknown or Not Reported | 3 | 4 | 3 | 10

OUTCOME MEASURES:

1. Primary Outcome: Systolic Blood Pressure
Description: Blood pressure measurements were taken by participants using a validated, WIFI-enabled blood pressure cuff manufactured by BlipCare and provided to study subjects prior to the baseline assessment. Measurements were automatically uploaded over a WIFI connection to the BlipHub app and study outcomes database. Participants followed a standardized measurement protocol based on the American Heart Association protocol for home blood pressure measurement, involving three consecutive measurements, taken one minute apart after a five-minute seated resting period. Measurements were not observed.
Time Frame: Baseline, 12 weeks, 24 weeks
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | BlipHub Mobile-web App | BlipHub Mobile-web App + Health Coaching | Usual Care
Number analyzed (Participants) | 67 | 68 | 68
mm Hg
  Baseline | 128.99 (12.77) | 131.4 (12.80) | 131.21 (12.82)
  12-week post-test | 127.45 (13.67) | 130.40 (14.40) | 130.00 (11.96)
  24-week follow-up | 127.50 (12.68) | 127.81 (12.31) | 128.90 (12.49)

2. Primary Outcome: Diastolic Blood Pressure
Description: as for outcome 1
Time Frame: Baseline, 12 weeks, 24 weeks
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | BlipHub Mobile-web App | BlipHub Mobile-web App + Health Coaching | Usual Care
Number analyzed (Participants) | 67 | 68 | 68
mm Hg
  Baseline | 76.95 (11.03) | 80.48 (10.10) | 77.83 (10.46)
  12-week post-test | 75.78 (10.42) | 76.80 (11.65) | 77.55 (11.15)
  24-week follow-up | 77.31 (11.60) | 78.11 (9.89) | 78.13 (9.46)

3. Primary Outcome: Body Weight
Description: Body weight measurements were taken by participants using a validated, WIFI-enabled weight scale manufactured by BlipCare and provided to study subjects prior to the baseline assessment. Measurements were automatically uploaded over a WIFI connection to the BlipHub app and study outcomes database. Participants were instructed to take weight measurements at the same time of day each time, preferably first thing in the morning after using the bathroom and before eating or drinking. The weight measurement taken on the date and time closest to the completion date and time of each individual's online survey for that assessment point was analyzed. If no measurements were available within two weeks on either side of that date, weight measurements were considered missing for that assessment period.
Time Frame: Baseline, 12 weeks, 24 weeks
Measure: Mean (Standard Deviation); unit: Pounds
Arm/Group | BlipHub Mobile-web App | BlipHub Mobile-web App + Health Coaching | Usual Care
Number analyzed (Participants) | 67 | 68 | 68
Pounds
  Baseline | 187.21 (49.67) | 196.65 (37.98) | 187.60 (48.76)
  12-week post-test | 187.61 (49.64) | 194.58 (38.60) | 194.05 (47.14)
  24-week follow-up | 187.67 (50.57) | 194.77 (39.00) | 196.60 (50.98)

4. Primary Outcome: Heart-healthy Dietary Intake (Number of Fruit/Vegetable Servings, White Meat Servings, Low-fat Dairy Servings)
Description: Participants were asked about their diet during the past month, using DASH-diet related items adapted from several validated food frequency questionnaires. Participants reported on servings consumed (e.g., never, 1-3 times last month, up to 5 or more times a day) of the following foods: fruits, vegetables, dairy, fats and meat. Number of servings was computed for heart-healthy foods (fruits, vegetables and lean meats).
Time Frame: Baseline, 12 weeks, 24 weeks
Measure: Mean (Standard Deviation); unit: Servings
Arm/Group | BlipHub Mobile-web App | BlipHub Mobile-web App + Health Coaching | Usual Care
Number analyzed (Participants) | 67 | 68 | 68
Servings
  Baseline | 5.98 (4.47) | 6.10 (4.74) | 5.85 (4.28)
  12-week post-test | 5.22 (3.71) | 6.22 (4.48) | 4.87 (3.93)
  24-week follow-up | 5.60 (4.32) | 6.03 (3.92) | 5.53 (4.25)

5. Primary Outcome: Heart-unhealthy Dietary Intake (Self-reported Number of Fat Servings, Red Meat Servings, Dairy Fat Servings)
Description: Participants were asked about their diet during the past month, using DASH-diet related items adapted from several validated food frequency questionnaires. Participants reported on servings consumed (e.g., never, 1-3 times last month, up to 5 or more times a day) of the following foods: fruits, vegetables, dairy, fats and meat. Number of servings was computed for heart-unhealthy foods (red, processed and high-fat prepared meats).
Time Frame: Baseline, 12 weeks, 24 weeks
Measure: Mean (Standard Deviation); unit: Servings
Arm/Group | BlipHub Mobile-web App | BlipHub Mobile-web App + Health Coaching | Usual Care
Number analyzed (Participants) | 67 | 68 | 68
Servings
  Baseline | 4.94 (4.72) | 4.54 (3.66) | 5.15 (3.62)
  12-week post-test | 4.33 (3.82) | 3.70 (2.61) | 4.12 (3.13)
  24-week follow-up | 4.17 (3.11) | 3.77 (3.80) | 4.61 (3.44)

6. Secondary Outcome: Self-reported Lifestyle Change Preparation Behaviors
Description: Participants were asked to self-report on days in the past two weeks in which they engaged in specific behaviors to prepare for or support healthy eating and physical activity (i.e., "preparation behaviors"). The scale comprised 15 items (e.g., thought about what you might do to try to lose weight) assessed on a 5-point scale (1=none (min), 5=12-14 days (max)). Mean score is reported, with higher scores indicating more frequent preparation behaviors. The scale showed good reliability (alpha=.91).
Time Frame: Baseline, 12 weeks, 24 weeks
Measure: Mean (Standard Deviation); unit: units on a Likert scale
Arm/Group | BlipHub Mobile-web App | BlipHub Mobile-web App + Health Coaching | Usual Care
Number analyzed (Participants) | 67 | 68 | 68
units on a Likert scale
  Baseline | 2.70 (0.89) | 2.52 (0.74) | 2.48 (0.88)
  12-week post-test | 2.78 (0.95) | 2.88 (0.84) | 2.48 (0.88)
  24-week follow-up | 2.67 (0.90) | 2.70 (0.85) | 2.45 (0.83)

7. Secondary Outcome: Self-reported Self-efficacy for Lifestyle Behaviors
Description: Five items assessed participants' confidence to engage in JNC-recommended healthy behaviors using a 5-item response option (1=not at all confident (min), 5=very confident (max)). Mean score is reported, with higher scores indicating higher self-efficacy. The scale showed good reliability (alpha=.79).
Time Frame: Baseline, 12 weeks, 24 weeks
Measure: Mean (Standard Deviation); unit: units on a Likert-type scale
Arm/Group | BlipHub Mobile-web App | BlipHub Mobile-web App + Health Coaching | Usual Care
Number analyzed (Participants) | 67 | 68 | 68
units on a Likert-type scale
  Baseline | 4.06 (0.60) | 4.10 (0.61) | 3.97 (0.73)
  12-week post-test | 3.67 (0.78) | 3.87 (0.60) | 3.65 (0.69)
  24-week follow-up | 3.71 (0.88) | 3.83 (0.61) | 3.70 (0.64)

ADVERSE EVENTS:
Time Frame: Adverse event monitoring lasted for 30 months, beginning with screening on 07/22/2013 and ending when the last participant completed the last blood pressure assessment on 3/25/2015.
Description: Blood pressure measurements (self-reported during screening and WIFI-transmitted for assessments) were monitored throughout data collection. Subjects with readings of systolic BP 160+ and/or diastolic BP 100+ were emailed with the recommendation to have their blood pressure checked by licensed healthcare professional.
Arm/Group | BlipHub Mobile-web App | BlipHub Mobile-web App + Health Coaching | Usual Care
Serious Adverse Events (participants affected / at risk) | 0/67 | 0/68 | 0/68
Other Adverse Events (participants affected / at risk) | 11/67 | 13/68 | 14/68
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BlipHub Mobile-web App (N=67) | BlipHub Mobile-web App + Health Coaching (N=68) | Usual Care (N=68)
Elevated BP (SBP 160+ or DBP 100+) (Vascular disorders) | 11 (11) | 13 (13) | 14 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes